CLINICAL TRIAL: NCT00383838
Title: Self-Selected Brief Alcohol Intervention for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21AA013284-01 (NIH)
Record Dates: First submitted 2006-03-20; First posted 2006-10-04 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2006-10

CONDITIONS: Alcohol Consumption; Drug Abuse
Keywords: brief motivational intervention; teens; substance use
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders

INTERVENTIONS:
Behavioral: brief, voluntary substance use intervention

SUMMARY:
Alcohol use among youth continues to be a major concern for this nation, with a large proportion of adolescents increasing their alcohol consumption as they transition from the 6th to the 8th grade. Although many adolescents experience alcohol-related problems, few actually seek help or treatment. This may be because traditional intervention approaches are not well suited for this age group. It is important to understand where adolescents turn to when they want to get help. The current project focuses on developing an alcohol intervention program for younger adolescents. We will conduct biannual surveys at two middle schools to assess alcohol and drug use patterns over three years. In years 2 and 3, we will implement an intervention in one of the schools.We will examine whether the intervention has an impact on subsequent alcohol use.

DETAILED DESCRIPTION:
Alcohol use among youth continues to be a major concern for this nation, with a large proportion of adolescents increasing their alcohol consumption as they transition from the 6th to the 8th grade. Although many adolescents experience alcohol-related problems, few actually seek help or treatment. This may be because traditional intervention approaches are not well suited for this age group. The aims of this project are to assess factors that impact younger adolescents' alcohol-related help-seeking behavior and to develop and standardize a developmentally sensitive self-change facilitation program. We will also preliminarily test the efficacy of the program in modifying the alcohol involvement (e.g., initiation, use, and problems) of middle school students. The focus of this grant is on younger adolescents (e.g., 12-15 years old), as they are particularly vulnerable to initiating alcohol use due to unique developmental issues. For example, peer conformity peaks during 6tn, 7th and 8th grade and declines thereafter. In addition, this age group is less likely to consider future consequences in the decision making process. Biannual surveys at two middle schools will assess alcohol and drug use patterns, help-seeking behavior and preferences, self-change efforts, and level of motivation for change. Year 1 data will be used to develop a voluntary brief intervention program that targets a variety of youth, including those who are just beginning to experiment with alcohol and those who may have experienced some problems due to their use. Primary objectives are: 1) to explore barriers and facilitative factors that promote/hinder younger adolescents' use of services, 2) use detailed survey information to design and pilot a self-change program, 3) examine alcohol involvement in relation to program utilization, and 4) preliminarily evaluate the efficacy of the intervention and overall patterns of service use. This study will extend facilitation of self-change research, as this program will be one of the first voluntary alcohol focused intervention programs to target middle school students.

ELIGIBILITY:
Inclusion Criteria:

* middle school student

Exclusion Criteria:

* none

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200
Dates: Start 2002-09; Study Completion 2005-06

PRIMARY OUTCOMES:
alcohol, tobacco, drug use
alcohol and drug consequences
self-change efforts
perceived peer use
positive and negative outcome expectancies
all measures taken biannually over a three year period

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J D'Amico, Ph.D., Principal Investigator — RAND